CLINICAL TRIAL: NCT03363373
Title: A Pivotal Phase 2 Trial of Antibody Naxitamab (hu3F8) and Granulocyte-Macrophage Colony Stimulating Factor (GM-CSF) in High-Risk Neuroblastoma Patients With Primary Refractory Disease or Incomplete Response to Salvage Treatment in Bone and/or Bone Marrow
Brief Title: Naxitamab for High-Risk Neuroblastoma Patients With Primary Refractory Disease or Incomplete Response to Salvage Treatment in Bone and/or Bone Marrow
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Y-mAbs Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201
Record Dates: First submitted 2017-11-06; First posted 2017-12-06 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Neuroblastoma
Keywords: Antibody, Neuroblastoma, Pediatric, Adult
MeSH Terms: conditions — Neuroblastoma | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; naxitamab

STUDY DESIGN:
Intervention Model Description: Patients will receive cycles of GM-CSF and Naxitamab every 4 weeks up to a total of 101 weeks. Safety and efficacy will be investigated with short-term follow-up at minimum 4 weeks after last treatment and with long-term follow-up for up to 3 years after end of treatment visit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- GM-CSF + Naxitamab (Experimental): Each investigational cycle is started with 5 days of GM-CSF administered at 250 µg/m2/day in advance of the start of Naxitamab administration. GM-CSF is thereafter administered at 500 µg/m2/day on days 1 to 5. As standard treatment, Naxitamab is administered at 3 mg/kg/day on days 1, 3, and 5 totalling 9 mg/kg per cycle. Treatment cycles are repeated every 4 weeks until CR or PR followed by 5 additional cycles every 4 weeks (±1 week). Subsequent cycles are repeated every 8 weeks (±2 weeks) through 101 weeks from first infusion at the discretion of the investigator. After end of treatment patients will enter a long-term follow up for up to 3 years after end of treatment visit.
  Interventions: Biological: GM-CSF + Naxitamab

INTERVENTIONS:
Biological: GM-CSF + Naxitamab — Granulocyte-Macrophage Colony Stimulating Factor (GM-CSF) and Humanized IgG1 monoclonal GD2 antibody

SUMMARY:
Children and adults diagnosed with high-risk neuroblastoma patients with primary refractory disease or incomplete response to salvage treatment in bone and/or bone marrow will be treated for up to 101 weeks with naxitamab and granulocyte-macrophage colony stimulating factor (GM-CSF). Patients will be followed for up to five years after first dose.

Naxitamab, also known as hu3F8 is a humanised monoclonal antibody targeting GD2

DETAILED DESCRIPTION:
Each patient will receive treatment for up to 101 weeks following the first Naxitamab administration. After the end of trial visit, each patient will enter a long-term follow-up where they will be monitored for up to 5 years after first treatment cycle.

Each investigational cycle is started with 5 days, days -4 to 0, of Granulocyte-Macrophage Colony Stimulating Factor (GM-CSF) administered at 250 µg/m2/day in advance of the start of Naxitamab administration. GM-CSF is thereafter administered at 500 µg/m2/day on days 1 to 5. As standard treatment, Naxitamab is administered at 3 mg/kg/day on days 1, 3, and 5, totalling 9 mg/kg per cycle.

Treatment cycles are repeated every 4 weeks (±1 week) until complete response or partial response followed by 5 additional cycles every 4 weeks (±1 week). Subsequent cycles are repeated every 8 weeks (±2 weeks) through 101 weeks from first infusion at the discretion of the investigator. End of treatment will take place around 8 weeks after the last cycle and thereafter long-term follow-up will continue.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of neuroblastoma as defined per International Neuroblastoma Response Criteria
* High-risk neuroblastoma patients with either primary refractory disease or incomplete response to salvage treatment (in both cases including stable disease, minor response and partial response) evaluable in bone and/or bone marrow.
* Life expectancy ≥ 6 months

Exclusion Criteria:

* Any systemic anti-cancer therapy, including chemotherapy or immunotherapy, within 3 weeks before 1st dose of GM-CSF
* Evaluable neuroblastoma outside bone and bone marrow
* Existing major organ dysfunction > Grade 2, with the exception of hearing loss, hematological status, kidney and liver function
* Active life-threatening infection

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2018-04-03 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Response rate during Naxitamab treatment | 101 weeks
  Overall objective response rate (ORR) during the Naxitamab treatment period that will be centrally assessed according to the International Neuroblastoma Response Criteria (INRC) modified with 123I-MIBG criteria and following the use of 18F FDG-PET for MIBG non-avid lesions.

SECONDARY OUTCOMES:
Incidence of adverse events and serious adverse events | 101 weeks
  Safety will be evaluated by the incidence of adverse events (AE) and serious adverse events (SAEs) graded according to CTCAE, version 4.0.
Duration of Response (DoR) | 101 weeks
  Length of time from patient response to disease progression.
Complete Response Rate | 101 weeks
  The complete response (CR) rate is defined as the fraction of patients experiencing a CR according to International Neuroblastoma Response Criteria (INRC) criteria during the treatment period.
Assessment of the maximum serum concentration (cmax) of naxitamab | Pre-naxitamab dose - 552 hours
  Calculation of maximum serum concentration of naxitamab will be calculated and summarized with descriptive statistics.
Assessment of the minimum serum concentration (cmin) of naxitamab | Pre-naxitamab dose - 552 hours
  Calculation of minimum serum concentration of naxitamab will be calculated and summarized with descriptive statistics.
Assessment of the clearance of naxitamab | Pre-naxitamab dose - 552 hours
  Calculation of clearance of naxitamab will be calculated and summarized with descriptive statistics.
Assessment of the volume of distribution of naxitamab | Pre-naxitamab dose - 552 hours
  Calculation of the volume of distribution of naxitamab will be calculated and summarized with descriptive statistics.
Assessment of the Area under the Curve (AUC) of naxitamab | Pre-naxitamab dose - 552 hours
  Calculation of the AUC of naxitamab will be calculated and summarized with descriptive statistics.
Assessment of the terminal half-life (t½) of naxitamab | Pre-naxitamab dose - 552 hours
  Calculation of the t½ of naxitamab will be calculated and summarized with descriptive statistics.
Assessment of anti-drug antibody (ADA) formation | Pre-naxitamab dose - 552 hours
  ADA formation will be investigated following a multi-tiered approach: A screening confirmation-titration analysis plus a ligand binding assay to examine a potential neutralizing effect of anti-naxitamab antibodies.
Intravenous (IV) opioid use (cycle 1) | 6 hours
  IV opioid use during cycle 1 defined as total dosage of IV morphine (or equivalent opioid) administered 2 hours before infusion until 4 hours after end of infusion of naxitamab
Intravenous (IV) opioid use (all cycles) | 101 weeks
  IV opioid use for each cycle during the trial defined as total dosage of IV morphine (or equivalent opioid) administered 2 hours before infusion until 4 hours after end of infusion of naxitamab
Hospitalization days (cycle 1) | 4 weeks
  Number of hospitalization days related to naxitamab during cycle 1, defined as number of overnight stays. Hospitalizations required solely for protocol-specified assessments (e.g., PK sampling) or non-medical circumstances are excluded
Safety of patients with positive human anti-drug antibody (ADA) | 101 weeks
  In patients with positive ADA at trial inclusion, safety will be evaluated by the incidence of AEs and SAEs graded according to CTCAE, version 4.0
Number of infusions done in an outpatient setting | 101 weeks
  Number of infusions done in an outpatient setting
Percentage of infusions done in an outpatient setting | 101 weeks
  Percentage of infusions done in an outpatient setting
Incidence of adverse events and serious adverse events in ADA positive patients | 101 weeks
  Safety will be evaluated by the incidence of adverse events (AE) and serious adverse events (SAEs) graded according to CTCAE, version 4.0 in ADA positive patients.
Progression Free Survival (PFS) | 5 years
  PFS, defined as the time from the first 1st infusion of naxitamab until progressive disease or death, whichever comes first
Overall Survival | 5 years
  The interval from the date of first dose of Naxitamab until the date of death due to any cause.
Happiness and activity levels | 39 days
  Happiness and activity levels will be measured over time and assessed by caretaker

CONTACTS AND LOCATIONS:
Locations (26):
- United States (6):
  - University of Florida, Gainesville, Florida
  - University of Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - M.D. Anderson Cancer Center, Houston, Texas
- The Hospital for Sick Children, Toronto, Canada
- Rigshospitalet, Copenhagen, Denmark
- Hopital pour enfants de la Timone, Marseille, Marseille, France
- Germany (3):
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - Johannes Gutenberg-Universität, Mainz
  - University Hospital Regensburg, Regensburg
- Hong Kong (2):
  - Hong Kong Children's Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Tata Memorial Centre, Mumbai, India
- Italy (3):
  - Giannina Gaslini Hospital, Genoa, Genoa
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Milan
  - Ospedale Pediatrico Bambino Gesù, Rome
- Spain (4):
  - Hospital Sant Joan de Déu, Barcelona
  - Hospital Infantil Universitario Niño Jesús, Madrid
  - Hospital Universitario Virgen Del Rocío, Seville
  - Hospital Universitario y Politécnico La Fe, Valencia
- United Kingdom (4):
  - The Royal Glasgow Children's Hospital, Glasgow
  - Leeds General Infirmary, Leeds
  - The Royal Marsden, London
  - University Hospital Southampton, Southampton

IPD SHARING:
Plan to Share IPD: Undecided